CLINICAL TRIAL: NCT05964946
Title: Real-life Study of the Characteristics of Patients Treated With Ilaris® (Canakinumab) for Gouty Arthritis in France
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CACZ885HFR01
Record Dates: First submitted 2023-07-20; First posted 2023-07-28 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Gouty Arthritis
MeSH Terms: conditions — Arthritis, Gouty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
This was a non-interventional, retrospective, cross-sectional, descriptive study, conducted on the National Health Data System (Système National des Données de Santé, SNDS).

The study did not modify the doctor-patient relationship, nor the management or follow-up of patients. Patients with dispensation of canakinumab for gouty arthritis were selected over the period from 08 April 2018 to 07 April 2020; index date was defined as date of the first dispensation of canakinumab in community pharmacy during study period.

Patients were described at index date. Medical history and comorbidities, and previous treatments for gouty arthritis were assessed during 3 years prior to index date. Co-treatments of interest for which standard treatments for gouty arthritis were contraindicated or required precautions for use were assessed during 6 months prior to index date.

ELIGIBILITY:
Inclusion Criteria:

* Received at least one reimbursement of Ilaris® from 08 April 2018 to 07 April 2020.
* Benefited from at least one of the following healthcare consumptions during 3 years prior to index date:

  o At least one hospitalization with a main diagnosis or a related diagnosis in a Medical Unit Summary or a significant associated diagnosis in a Standardized Discharge Summary corresponding to the International Classification of Diseases, 10th Revision (ICD-10) code:
  * M10.0 "Idiopathic gout"
  * M10.1 "Saturnine gout"
  * M10.2 "Medicated gout"
  * M10.3 "Gout due to impaired renal function"
  * M10.4 "Other secondary gout"
  * M10.9 "Gout, unspecified"
* And/or an active long-term disease (Affection Longue Durée, ALD) with an ICD-10 code: "M10 Gout"
* And/or at least one dispensation of colchicine and urate-lowering therapy (allopurinol and/or febuxostat and/or benzbromarone and/or probenecid) at any time.

Exclusion Criteria:

None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This was a retrospective, noninterventional cohort study.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2020-06-24 (Actual); Primary Completion 2022-07-29 (Actual); Study Completion 2022-07-29 (Actual)

PRIMARY OUTCOMES:
Number of patients treated with canakinumab in France for the treatment of gouty arthritis | 2 years

SECONDARY OUTCOMES:
Mean age of patients | 3 years
Number of male patients | 3 years
Geographic location of patients | 3 years
Number of patients with previous treatments for gouty arthritis | 3 years
Medical history of patients | 3 years
Number of patients with comorbidities | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis, Paris, France